CLINICAL TRIAL: NCT02045108
Title: Modifying Alcohol Approach Motivations With tDCS and Cognitive Retraining
Brief Title: Cognitive Retraining and Brain Stimulation for Alcohol Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Mind Research Network (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 20-520; 1R21AA021201-01A1 (NIH)
Record Dates: First submitted 2014-01-20; First posted 2014-01-24 (Estimated); Results first posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Binge Drinking
MeSH Terms: conditions — Binge Drinking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Active TDCS + Active Retraining (Experimental): 2.0 milliamps (mA) of TDCS applied during active alcohol avoidance retraining
  Interventions: Behavioral: Active Retraining; Device: Active TDCS
- Sham TDCS + Active Retraining (Experimental): .1 mA of TDCS applied during active alcohol avoidance retraining
  Interventions: Behavioral: Active Retraining; Device: Sham TDCS
- Active TDCS + Sham retraining (Experimental): 2.0 mA of TDCS applied during sham alcohol avoidance retraining
  Interventions: Device: Active TDCS; Behavioral: Sham Retraining
- Sham TDCS + Sham Retraining (Sham Comparator): 0.1 mA of TDCS applied during sham alcohol avoidance retraining
  Interventions: Device: Sham TDCS; Behavioral: Sham Retraining

INTERVENTIONS:
Behavioral: Active Retraining
  Arms: Active TDCS + Active Retraining; Sham TDCS + Active Retraining
Device: Sham TDCS
  Arms: Sham TDCS + Active Retraining; Sham TDCS + Sham Retraining
Device: Active TDCS
  Arms: Active TDCS + Active Retraining; Active TDCS + Sham retraining
Behavioral: Sham Retraining
  Arms: Active TDCS + Sham retraining; Sham TDCS + Sham Retraining

SUMMARY:
The overarching goal of this study is to determine whether combined cognitive training and Transcranial Direct Current Stimulation (tDCS) reduces drinking in high-risk drinkers. To this end, specific study purposes are: 1) replicate previous findings that cognitive retraining reduces drinking levels, 2) test whether cognitive retraining can be enhanced with tDCS, and 3) investigate the neural changes that result from cognitive retraining and tDCS. We hypothesize that those participants who receive alcohol avoidance cognitive training will have greater reductions in drinking. In turn, those participants who receive a higher level of applied tDCS during alcohol avoidance response training will have better avoidance learning, as well as, a larger reduction in drinking behavior. Finally, those participants receiving a higher level of applied tDCS will have more neuronal response associated with alcohol avoidance during the brain imaging session.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-30 years
* At least five binge drinking episodes (4+ drinks for men; 3+ drinks for women) for the past month
* Alcohol Use Disorder Identification Test (AUDIT) score greater than 8
* Right handed

Exclusion Criteria:

* History of treatment for alcohol dependence (AD) or desire for treatment
* History of alcohol withdrawal
* History of brain injury
* Currently taking psychotropic medications (e.g. antidepressants, antipsychotics)
* Female subjects who are pregnant
* Evidence of recent illicit drug use on a urine screen
* Left handed
* Prior participation in a brain stimulation study
* Implanted brain medical devices
* Electromedical devices
* Latex allergy

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric D Claus, Ph.D., Principal Investigator — Mind Research Network and LBERI
Locations (1):
- The Mind Research Network and University of New Mexico Center on Alcoholism, Substance Abuse and Addiction, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Active TDCS + Active Retraining: 2.0 milliamps (mA) of transcranial direct current stimulation (TDCS) applied during active alcohol avoidance retraining
  Active Retraining
  Active TDCS
- Sham TDCS + Active Retraining: .1 mA of TDCS applied during active alcohol avoidance retraining
  Active Retraining
  Sham TDCS
- Active TDCS + Sham Retraining: 2.0 mA of TDCS applied during sham alcohol avoidance retraining
  Active TDCS
  Sham Retraining
- Sham TDCS + Sham Retraining: 0.1 mA of TDCS applied during sham alcohol avoidance retraining
  Sham TDCS
  Sham Retraining
Period: Overall Study
Arm/Group | Active TDCS + Active Retraining | Sham TDCS + Active Retraining | Active TDCS + Sham Retraining | Sham TDCS + Sham Retraining
Started | 22 | 15 | 20 | 20
Completed | 21 | 12 | 18 | 19
Not Completed | 1 | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Active TDCS + Active Retraining: 2.0 milliamps (mA) of TDCS applied during active alcohol avoidance retraining
  Active Retraining
  Active TDCS
- Total: Total of all reporting groups
Arm/Group | Active TDCS + Active Retraining | Sham TDCS + Active Retraining | Active TDCS + Sham Retraining | Sham TDCS + Sham Retraining | Total
Number analyzed (Participants) | 22 | 15 | 20 | 20 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.50 (2.70) | 24.80 (2.78) | 24.95 (2.80) | 22.90 (1.92) | 24.55 (2.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 6 | 6 | 24
  Male | 14 | 11 | 14 | 14 | 53

OUTCOME MEASURES:

1. Primary Outcome: Drinks Per Drinking Day
Description: Number of standard drinks will be assessed using the Timeline Follow-back method to obtain the number of drinks consumed on each day of the prior 30 days. Drinks per drinking day will be the mean number of drinks consumed on days on which alcohol was consumed.
Time Frame: Screening Visit
Population: At-risk alcohol drinkers ages 21-30
Measure: Mean (Standard Deviation); unit: drinks per drinking day
Arm/Group | Active TDCS + Active Retraining | Sham TDCS + Active Retraining | Active TDCS + Sham Retraining | Sham TDCS + Sham Retraining
Number analyzed (Participants) | 22 | 15 | 20 | 20
drinks per drinking day | 6.1 (4.1) | 6.8 (3.4) | 6.6 (3.3) | 7.5 (3.4)

2. Primary Outcome: Alcohol Approach Bias
Description: For each participant, bias is computed by taking the median response times to approaching alcohol pictures - response times to avoiding alcohol pictures, as measured with a pull or push of a joystick. Group means of these medians are presented as the outcome measure.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Active TDCS + Active Retraining | Sham TDCS + Active Retraining | Active TDCS + Sham Retraining | Sham TDCS + Sham Retraining
Number analyzed (Participants) | 22 | 15 | 20 | 20
milliseconds | 6.0 (84.6) | 17.4 (114.9) | 26.4 (110.0) | 20.3 (111.9)

3. Primary Outcome: Drinks Per Drinking Day
Description: Number of standard drinks will be assessed using the Timeline Follow-back method to obtain the number of drinks consumed on each day since the last administration of the Timeline Follow-back. Drinks per drinking day will be the mean number of drinks consumed on days on which alcohol was consumed.
Time Frame: 1 week post-baseline
Measure: Mean (Standard Deviation); unit: standard drinks per drinking day
Arm/Group | Active TDCS + Active Retraining | Sham TDCS + Active Retraining | Active TDCS + Sham Retraining | Sham TDCS + Sham Retraining
Number analyzed (Participants) | 22 | 15 | 20 | 20
standard drinks per drinking day | 4.7 (2.6) | 6.1 (2.8) | 5.2 (2.6) | 4.8 (2.7)

4. Primary Outcome: Drinks Per Drinking Day
Description: as for outcome 3
Time Frame: 2 weeks post-baseline
Population: Two participants in the Active TDCS/Sham retraining and one participant in the Sham TDCS/Active Retraining condition failed to show up for this appointment and therefore were not included in the summary data.
Measure: Mean (Standard Deviation); unit: standard drinks
Arm/Group | Active TDCS + Active Retraining | Sham TDCS + Active Retraining | Active TDCS + Sham Retraining | Sham TDCS + Sham Retraining
Number analyzed (Participants) | 22 | 14 | 18 | 20
standard drinks | 5.1 (2.2) | 6.0 (2.8) | 6.5 (3.5) | 4.6 (2.0)

5. Primary Outcome: Drinks Per Drinking Day
Description: as for outcome 3
Time Frame: 3 weeks post-baseline
Population: Two participant in the Sham TDCS/Active Retraining, two participants in the Active TDCS/Sham retraining, and one participants in the Sham TDCS/Active Retraining condition failed to show up for this appointment and therefore were not included in the summary data.
Measure: Mean (Standard Deviation); unit: standard drinks
Arm/Group | Active TDCS + Active Retraining | Sham TDCS + Active Retraining | Active TDCS + Sham Retraining | Sham TDCS + Sham Retraining
Number analyzed (Participants) | 22 | 13 | 18 | 19
standard drinks | 5.8 (5.1) | 5.5 (2.7) | 5.5 (2.7) | 5.0 (5.3)

6. Primary Outcome: Drinks Per Drinking Day
Description: as for outcome 3
Time Frame: 4 weeks post-baseline
Population: One participant in the Active TDCS/Active Retraining, three participants in the Sham TDCS/Active Retraining, two participants in the Active TDCS/Sham retraining, and one participant in the Sham TDCS/Active Retraining condition failed to show up for this appointment and therefore were not included in the summary data.
Measure: Mean (Standard Deviation); unit: standard drinks
Arm/Group | Active TDCS + Active Retraining | Sham TDCS + Active Retraining | Active TDCS + Sham Retraining | Sham TDCS + Sham Retraining
Number analyzed (Participants) | 21 | 12 | 18 | 19
standard drinks | 4.9 (2.9) | 7.5 (3.4) | 5.2 (4.3) | 5.2 (2.2)

7. Primary Outcome: Drinks Per Drinking Day
Description: as for outcome 3
Time Frame: 5 weeks post-baseline
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: standard drinks
Arm/Group | Active TDCS + Active Retraining | Sham TDCS + Active Retraining | Active TDCS + Sham Retraining | Sham TDCS + Sham Retraining
Number analyzed (Participants) | 21 | 12 | 18 | 19
standard drinks | 5.7 (1.9) | 6.5 (4.4) | 5.9 (3.7) | 5.1 (3.5)

8. Primary Outcome: Drinks Per Drinking Day
Description: as for outcome 3
Time Frame: 8 weeks post-baseline
Population: Two participants in the Active TDCS/Active Retraining, four participants in the Sham TDCS/Active Retraining, two participants in the Active TDCS/Sham retraining, and three participants in the Sham TDCS/Active Retraining condition failed to show up for this appointment and therefore were not included in the summary data.
Measure: Mean (Standard Deviation); unit: standard drinks
Arm/Group | Active TDCS + Active Retraining | Sham TDCS + Active Retraining | Active TDCS + Sham Retraining | Sham TDCS + Sham Retraining
Number analyzed (Participants) | 20 | 11 | 18 | 17
standard drinks | 4.5 (2.5) | 6.6 (2.7) | 5.7 (3.1) | 5.5 (2.2)

9. Primary Outcome: Alcohol Approach Bias
Description: as for outcome 2
Time Frame: 1 week after treatment
Population: Three participants in the Sham TDCS/Active Retraining, one participant in the Active TDCS/Sham retraining, and one participant in the Sham TDCS/Active Retraining condition failed to show up for this appointment and therefore were not included in the summary data.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Active TDCS + Active Retraining | Sham TDCS + Active Retraining | Active TDCS + Sham Retraining | Sham TDCS + Sham Retraining
Number analyzed (Participants) | 22 | 12 | 19 | 19
milliseconds | 41.6 (87.6) | 143.6 (219.8) | 51.9 (85.3) | 66.6 (102.6)

10. Primary Outcome: Drinks Per Drinking Day
Description: as for outcome 3
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: drinks per drinking day
Arm/Group | Active TDCS + Active Retraining | Sham TDCS + Active Retraining | Active TDCS + Sham Retraining | Sham TDCS + Sham Retraining
Number analyzed (Participants) | 22 | 15 | 20 | 20
drinks per drinking day | 5.7 (1.9) | 5.5 (2.9) | 6.2 (3.6) | 6.1 (4.0)

ADVERSE EVENTS:
Arm/Group | Active TDCS + Active Retraining | Sham TDCS + Active Retraining | Active TDCS + Sham Retraining | Sham TDCS + Sham Retraining
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/15 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/15 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/22 | 1/15 | 1/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TDCS + Active Retraining (N=22) | Sham TDCS + Active Retraining (N=15) | Active TDCS + Sham Retraining (N=20) | Sham TDCS + Sham Retraining (N=20)
Redness at stimulation site (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No